CLINICAL TRIAL: NCT03759808
Title: Cognitive Behavioral Treatment for Patients With Chronic Post-Concussion Symptoms
Brief Title: Treatment for Patients With Chronic Post-Concussion Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Robert F. Asarnow, Ph.D, Study Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-000346
Record Dates: First submitted 2018-09-20; First posted 2018-11-30 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Mild Traumatic Brain Injury; Concussion Post Syndrome
Keywords: post-concussion syndrome; mild traumatic brain injury; autonomic dysfunction; concussion; capnometry-assisted respiratory training; cognitive behavioral therapy
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome; Primary Dysautonomias | interventions — Psychosocial Intervention

STUDY DESIGN:
Intervention Model Description: An open trial will be conducted in patients with persistent post-concussion symptoms compared to non-injured controls in order to determine whether the intervention (controlled breathing and cognitive behavioral therapy for anxiety) improves parasympathetic, HPA axis activity and cerebral blood flow, and whether improvement in parasympathetic and HPA axis activity predicts reduction in PPCS symptoms. We will compare baseline evaluations to the evaluation conducted after brief CBT and controlled breathing training to demonstrate the feasibility of normalizing parasympathetic, and HPA axis activity via this intervention. If we obtain the predicted results in the current study we will design a much larger study to identify the mechanisms of change. Healthy, non-injured control participants will provide normative data on all measures except for concussion-relevant outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Persistent Post-Concussion Symptoms (Experimental): Concussed participants with persistent post-concussion symptoms (PPCS) who receive the psychological intervention.
  Interventions: Behavioral: Psychological Intervention

INTERVENTIONS:
Behavioral: Psychological Intervention — Psychological treatment protocol designed to treat anxiety and avoidance in an adolescent/young adult population. The focus of treatment will be to address cognitive and behavioral factors associated with prolonged symptoms. Cognitive factors that may be addressed include, but are not limited to, catastrophizing, black or white thinking, and false expectations. Behavior factors that may be addressed include, but are not limited to, avoidance, relaxation, and behavioral activation. The psychological intervention is also designed to help reduce psychophysiological arousal associated with anxiety and stress. Participants will also be taught controlled shallow breathing exercises designed to normalize the ratio of sympathetic/parasympathetic activity.

SUMMARY:
The current project will examine the effect of a brief psychological intervention on post-concussion symptoms, neurocognitive function, cerebral blood flow (CBF), and psychophysiological and salivary cortisol markers of autonomic nervous system (ANS) in a sample of 20 participants between 13-25 years of age who experience long-term post-concussive (PC) symptoms 2-9 months post-injury as well as 20 age- and sex-matched controls (non-injured) participants to provide normative data on all the above measures except for concussive symptoms.

DETAILED DESCRIPTION:
Participants with concussion will participate in six, home-based interventions designed to treat cognitive-behavioral factors that are maintaining their symptoms. The investigators hypothesize that the prolonged PC symptoms are in part due to disruption of autonomic nervous system function post-injury as well as exacerbation by the psychological response to the injury. This hypothesis is based on evidence showing that PC symptoms, including headache, fatigue, dizziness, and heightened anxiety overlap with upregulated sympathetic activity and elevated levels of salivary cortisol. There is evidence linking cognitive-behavioral factors (e.g., catastrophizing) to prolonged symptoms of autonomic overactivation after injury (e.g., anxiety, pain, etc.). The participants are taught shallow breathing techniques to normalize parasympathetic activity and provide cognitive-behavioral treatment to reduce psychological reactions to the injury that exacerbate the autonomic disruption and prolong recovery.

ELIGIBILITY:
Inclusion criteria for patients:

* Between the ages of 13-25
* Diagnosed with a concussion or mild traumatic brain injury by a physician
* Currently experiencing post-concussive symptoms for at least two months after their injury but no longer than 9 months.
* Fluent English speaker

Exclusion Criteria:

* History of/or comorbid neurological conditions that might affect performance (including history of stroke, seizure disorder, moderate to severe traumatic brain injury, anoxia)
* Severe cardiovascular conditions.
* History of psychosis and current substance abuse or dependence.
* Current severe symptoms of depression and/or anxiety.

Additional Exclusion Criteria for Controls:

* No history of concussion in the past year.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Self-Reported Symptoms After Treatment | baseline and 6 weeks
  Severity of self-reported symptoms on the Post-Concussion Symptom Inventory
Change Self-Reported Quality of Life After Treatment | baseline and 6 weeks
  Self-reported scores on quality of life on Global Quality of Life Scale

SECONDARY OUTCOMES:
Change in cerebral blood flow stress after treatment | baseline and 6 weeks
  Changes in cerebral blood flow dynamics in bilateral middle cerebral arteries as measured by transcranial doppler.
Change in peak salivary cortisol after treatment | baseline and 6 weeks
  Changes in peak salivary cortisol concentration will be measured in response to stress paradigm. Measurements will be taken just prior to stress paradigm and then 20 minutes after its conclusion.
Change in respiration rate after treatment | baseline and 6 weeks
  Changes in respiration rate as measured through capnometer in response to stress paradigm
Change in end-tidal carbon dioxide after treatment | baseline and 6 weeks
  Changes in end-tidal carbon dioxide measurement in response to stress paradigm measured through capnometer in mmHg
Change in heart rate after treatment | baseline and 6 weeks
  Changes in heart rate (beats per minute) in response to stress paradigm measured through Biopac system.
Change in blood pressure after treatment | baseline and 6 weeks
  Changes in blood pressure (systolic/dyastolic in mmHg) in response to stress paradigm measured through Biopac system.

OTHER OUTCOMES:
Change in depressive symptoms after treatment | baseline and 6 weeks
  Self-report measure of cognitive and somatic symptoms of depression, Beck Depression Inventory (BDI-II)
Change in anxiety symptoms after treatment | baseline and 6 weeks
  Self-report measure of cognitive and somatic symptoms of anxiety, Beck Anxiety Inventory (BAI)
Change in sleep quality after treatment | baseline and 6 weeks
  Self-report measure of sleep dysfunction, Pittsburgh Sleep Quality Index (PSQI)
Change in neurocognitive performance after treatment | baseline and 6 weeks
  Selected subtest performance on attention, learning and memory, processing speed, and verbal fluency as measured by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) standardized assessment.
Change in perceived cognitive exertion after treatment | baseline and 6 weeks
  Change in self-reported physical, emotional, and perceived cognitive symptoms from pre- to post-neurocognitive assessment.
Change in illness perception after treatment | baseline and 6 weeks
  Change in self-reported perception of illness as measured by the Brief Illness Perception Questionnaire.
Change in behavioral avoidance and distress after treatment | baseline and 6 weeks
  Change in self-reported behavioral avoidance and distress due to anxiety as measured by the UCLA Behavioral Avoidance and Distress Scale
Change in disability perception due to injury after treatment | baseline and 6 weeks
  Change in self-reported disability in social, occupational, and family/home functioning as measured by the Sheehan Disability Scale
Change in orthostatic blood pressure after treatment | baseline and 6 weeks
  Change in orthostatic blood pressure obtained via measurements in three different positions: supine, upright sitting, and standing, each held for 5 minutes. Measurement obtained via Biopac double finger cuff.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Asarnow, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication will be shared if requested by other researchers. These data will include Study Protocol, Statistical Analysis Plan, and Clinical Study Report. Data will be made available for sharing 6 months after publication and be available for a time frame of 2 years following initial publication. Access to IPD will be considered for researchers with a graduate degree or above for post-hoc analyses or replication efforts. Applications to access individual participant data will be reviewed by principal investigator and appointed co-investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months following initial publication, lasting for 2 years after initial publication.
Access Criteria: Access to individual participant data will be considered for researchers with a graduate degree or above for post-hoc analyses or replication efforts. Applications to access individual participant data will be reviewed by principal investigator and appointed co-investigators.